CLINICAL TRIAL: NCT01758952
Title: Multi-center Prospective Investigation of Incidence and Risk Factors of Peri-operative Stroke in Non-cardiac,Non-neurosurgical Surgeries and Practicability of NIHSS in Screening Peri-operative Strokes
Brief Title: Incidence and Risk Factors of Peri-operative Stroke in Non-cardiac,Non-neurosurgical Surgeries
Acronym: POSIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: Peri-operativeStroke
Record Dates: First submitted 2012-12-23; First posted 2013-01-01 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2013-11

CONDITIONS: Peri-operative Stroke; Perioperative Adverse Events; Non-cardiac Surgery; Non-neurosurgical Surgery
Keywords: Peri-operative stroke; incidence; risk factors; prospective

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Beijing Chaoyang Hospital: 2000 cases
- Peking University Hospital: 2000 cases
- Zhongshan Hospital of Fudan University: 2000 cases
- Tongji Hospital, Wuhan: 2000 cases
- Tangdu Hospital, Xi'an: 2000 cases
- The Prince Welsh Hospital: 1000 cases

SUMMARY:
Stroke is an important cause of perioperative morbidity and mortality, particularly in patients > 60 years. In cardiac, neurological and carotid surgery the incidence is known to be high (2.2-5.2%). However, little is known regarding perioperative stroke following other types of surgery including general, urological, orthopedic, thoracic and gynecological procedures. We therefore propose to undertake a multicenter, observational cohort study, to determine the current incidence of, the risk factors for, and outcome associated with perioperative stroke in patients undergoing non-cardiac and non-neurological surgery.

DETAILED DESCRIPTION:
Patient population: Prospective cohort study of 10,000 adults undergoing non-cardiac, non-neurological surgery.

Screening and enrollment: Consecutive patients undergoing (elective or emergency) non-cardiac, non-neurosurgical surgeries will be recruited.

Monitoring, follow-up, and data collection: Usual treatment will be provided. Demographic details will be recorded. Patients will be visited regularly in hospital. Patient will be reviewed for neurologic deficit using the mNIHSS. Brain imaging will be performed to confirm stroke event. Follow-up at 30 days after discharge will be done to ascertain if there is any adverse outcome.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 60 Years and older
* Genders Eligible for Study: Both
* Accepts Healthy Volunteers: No
* Sampling Method: Probability Sample

Exclusion Criteria:

* hospital stay after surgery less than 3 days
* not consent of the assessment
* surgery canceled

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We propose a sample size of 10,000 patients to ensure a stable logistic model for an anticipated stroke rate of 1.0%.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
perioperative stroke occurs during and within 30 days after surgery. | 30 days after suegery
  The primary outcome is perioperative stroke occurs during and within 30 days after surgery. This is defined as cerebral infarction or hemorrhage on computer tomography or magnetic resonance scan, or new neurological signs (paralysis, weakness or speech difficulties) lasting more than 24 hours or leading to death. The mechanism of stroke will be classified using the Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria.

SECONDARY OUTCOMES:
total mortality and other major vascular complications up until 30 days after surgery | 30 days after suegery
  Secondary outcomes include total mortality and other major vascular complications up until 30 days after surgery:
  1. Myocardial infarction is defined according to recent universal definition of myocardial infarction;
  2. Nonfatal cardiac arrest is a successful resuscitation from either documented or presumed ventricular fibrillation or sustained ventricular tachycardia or asystole;
  3. Pulmonary embolism;
  4. Congestive heart failure is defined by both clinical and radiographic evidence;
  5. Clinically significant atrial fibrillation is defined as atrial fibrillation that results in angina, congestive heart failure, symptomatic hypotension, or that requires treatment with a rate controlling drug, antiarrhythmic drug, or electrical cardioversion;
  6. Cardiac death: defined as any death with a cardiovascular cause, including deaths following a cardiovascular procedure, cardiac arrest, myocardial infarction, pulmonary embolus, stroke, hemorrhage, or deaths due to unknown cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Yue, MD, Study Chair — Beijing Chao Yang Hospital
Locations (6):
- China (6):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - No.1 Hospital of Peking University, Beijing
  - Prince of Wales Hospital, Hong Kong
  - Zhongshan Hospital, Fudan University, Shanghai
  - Tongji Hospital, Huazhong University of Science and Technology, Wuhan
  - Tangdu Hospital, The Fourth Military Medical University, Xi'an

REFERENCES:
- [Background] Ng JL, Chan MT, Gelb AW. Perioperative stroke in noncardiac, nonneurosurgical surgery. Anesthesiology. 2011 Oct;115(4):879-90. doi: 10.1097/ALN.0b013e31822e9499. PMID 21862923